CLINICAL TRIAL: NCT01903148
Title: ANEMIA MANAGEMENT IN CHRONIC KIDNEY DISEASE NOT ON DIALYSIS PATIENTS AFTER THE ERBP WORKING GROUP RECOMMENDATIONS
Brief Title: Anemia Management in Chronic Kidney Disease Not on Dialysis Patients After the European Renal Best Practice (ERBP) Working Group Recommendations
Acronym: ACERCA
Status: Completed | Type: Observational
Sponsor: Fundación Senefro (Other)
Responsible Party: Sponsor
Other Study IDs: SEN-AEE-2011-01
Record Dates: First submitted 2013-07-12; First posted 2013-07-19 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-11

CONDITIONS: ANEMIA
Keywords: ANEMIA IN CHRONIC KIDNEY DISEASE PATIENTS NOT ON DIALYSIS
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the impact of the last recommendations of the European Anemia Working Group ERBP in the anemia management in the achievement of the therapeutic goal of Hb 11-12 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with anemia secondary to chronic kidney disease (CKD) not on dialysis.
* Patients starting anemia treatment (naïve) after six months of the last recommendations of the European Anemia Working Group ERBP (January 2011).
* Patients in treatment who changed from previous ESA treatment since January 2011 (converted patients

Exclusion Criteria:

* Patients in Erythropoiesis Stimulating Agents (ESA) dose adjustment period.
* Kidney transplant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with anemia secondary to chronic kidney disease (CKD) not on dyalisis.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Martinez Castelao, Doctor, Principal Investigator — Hospital Bellvitge; Aleix Cases, Doctor, Principal Investigator — Hospital Clinic of Barcelona
Locations (29):
- Spain (29):
  - Hospital Puerto Real, Cadiz, Andalusia
  - Hospital de Jerez, Jerez de la Frontera, Andalusia
  - Clínico V. Victoria, Málaga, Andalusia
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Nuestra Señora De Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital Virgen de la Luz, Toledo, Castille-La Mancha
  - Fundación Puigvert, Barcelona, Catalonia
  - Hospital Bellvige, Barcelona, Catalonia
  - Hospital Bellvitge, Barcelona, Catalonia
  - Hospital Clinic, Barcelona, Catalonia
  - Hospital Germans Trias i Pujol, Barcelona, Catalonia
  - Hospital Valld'Hebron, Barcelona, Catalonia
  - Sagrat Cor, Barcelona, Catalonia
  - Clinica Girona, Girona, Catalonia
  - Hospital Josep Trueta, Girona, Catalonia
  - Arquitecto Marcide, Ferrol, Galicia
  - Complexo Hospitalario de Ourense, Ourense, Galicia
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital General de Alicante, Alicante, Valencia
  - Hospital de Castellón, Castellon, Valencia
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Dr. Peset, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nephrology Units of 30 Spanish hospitals.
Pre-assignment Details: 14 patients were excluded because they didn't fulfill the eligibility criteria
Groups:
- Patients With Anemia and CKD: Adults patients with anemia secondary to chronic kidney disease (CKD) not on dialysis.
Period: Overall Study
Arm/Group | Patients With Anemia and CKD
Started | 441
Completed | 441
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Converted Patients: Patients in treatment who changed from previous ESA treatment since January 2011
- Naïve Patients: Patients starting anemia treatment (naïve) after six months of the last recommendations of the Anemia Working Group of ERBP (January 2011)
- Total: Total of all reporting groups
Arm/Group | Converted Patients | Naïve Patients | Total
Number analyzed (Participants) | 143 | 298 | 441
Age Continuous [Mean (Standard Deviation); unit: years] | 73.5 (13.9) | 72.9 (12.5) | 73.1 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 152 | 229
  Male | 66 | 146 | 212

OUTCOME MEASURES:

1. Primary Outcome: % Patients Achieving Target Hemoglobin Levels
Description: % patients with Hb levels between 11-12 mg/dl
Time Frame: 1 day because is a crosssectional study with only a visit
Measure: Number; unit: percentage of participants
Arm/Group | Converted Patients | Naïve Patients
Number analyzed (Participants) | 143 | 298
percentage of participants | 42.5 (1.3) | 35.3 (1.3)

2. Secondary Outcome: Hemoglobin Levels Per Type of Patients
Description: levels Hb and type of patients
Time Frame: 1 day
Population: n represents the number of participants analyzed for each category respectively (converted patients, naïve patients)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Converted Patients | Naïve Patients
Number analyzed (Participants) | 143 | 298
mg/dl
  Hb levels in non diabetics patients, n=79, 163 | 11.6 (1.2) | 11.5 (1.2)
  Hb levels in diabetics patients, n=64, 135 | 11.4 (1.3) | 11.1 (1.3)
  Hb levels patients non cardiovasdisease, n=76, 151 | 11.4 (1.2) | 11.5 (1.3)
  Hb levels patients cardiovasculardisease, n=67,147 | 11.7 (1.4) | 11.2 (1.2)
  Hb levels patients noncerebrovadisease, n=125, 265 | 11.6 (1.2) | 11.3 (1.3)
  Hb levels patients with cerebrovadisease n=18, 33 | 11.4 (1.7) | 11.4 (1.1)
  Hb levels patients non cancer, n=129,257 | 11.5 (1.3) | 11.3 (1.3)
  Hb levels patients with cancer n=14, 41 | 11.6 (1.2) | 11.3 (1.2)

3. Secondary Outcome: Patients With Hb>12
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Converted Patients | Naïve Patients
Number analyzed (Participants) | 143 | 298
participants | 52 | 71

4. Secondary Outcome: % Patients With Erythropoiesis Stimulating Agents (ESA) Therapy
Description: know the treatments ESA for maintenance of hb levels
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Converted Patients | Naïve Patients
Number analyzed (Participants) | 143 | 298
percentage of participants
  Mircera | 74.1 | 83.4
  Darbepoetin | 19.6 | 13.1
  Epoetin alfa | 2.1 | 1.7
  Epoetin beta | 4.2 | 1.7

5. Secondary Outcome: Iron Treatment
Description: Patients with supplementary Iron treatment to ESA
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Converted Patients | Naïve Patients
Number analyzed (Participants) | 143 | 298
participants | 68 | 175

6. Secondary Outcome: Patients With Hb<11
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Converted Patients | Naïve Patients
Number analyzed (Participants) | 143 | 298
participants | 38 | 98

ADVERSE EVENTS:
Arm/Group | Converted Patients | Naïve Patients
Serious Adverse Events (participants affected / at risk) | 1/143 | 1/298
Other Adverse Events (participants affected / at risk) | 3/143 | 1/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Converted Patients (N=143) | Naïve Patients (N=298)
Hipercalcemia (Vascular disorders) | 1 (1) | 0 (0)
Cardiac insufficiency left side (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Converted Patients (N=143) | Naïve Patients (N=298)
Precordial pain (Cardiac disorders) | 1 (1) | 0 (0)
auricular fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Urinary infection (Renal and urinary disorders) | 1 (1) | 0 (0)
orquiepididimitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Change sounds nefrostomia (Renal and urinary disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less